CLINICAL TRIAL: NCT05100108
Title: Effects of a Dog-assisted Therapy on Quality of Life, Work Engagement and Burnout Among Professionals Working in a School for Special Education
Brief Title: A Dog-assisted Therapy to Reduce Burnout Among Professionals Working in a School for Special Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daniel Collado-Mateo (Other)
Collaborators: Asociación Dame La Pata (Unknown)
Responsible Party: Sponsor-Investigator, Daniel Collado-Mateo, Assistant Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAI_Teachers
Record Dates: First submitted 2021-10-16; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Occupational Groups; Work Related Stress
Keywords: dog-assisted; Burnout; Quality of life; Work Engagement; Human-animal interaction; Animal-assisted
MeSH Terms: conditions — Occupational Stress; Burnout, Psychological; Human-Animal Interaction | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two groups: a) the experimental group and b) a control group (waiting list)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be aware of the group they belong. Assessors and investigators will not be aware of the group participants belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): They will be on a waiting list. They will be assessed before and after the 8 week program but will not take part in it.
- Experimental group (Experimental): Participants in this group will take part in the 8 sessions of dog-assisted therapy. They will be assessed before and after the 8 week program.
  Interventions: Behavioral: Dog-assisted therapy

INTERVENTIONS:
Behavioral: Dog-assisted therapy — The program will involve 8 sessions, conducted once a week for 8 weeks. Each session will include three parts: 1) a welcome part aimed to get in touch with the dog, 2) a main part, where participants will be taught basic notions about dog training and then try to train the dogs. In this part, the patients will perform different activities and exercises with the dog. 3) A closing part to relaxation and say goodbye to the dogs.
  Other Names: animal-assisted therapy; animal-assisted intervention
  Arms: Experimental group

SUMMARY:
This randomized controlled trial aims to evaluate the effects of an 8-week program consisting of dog-assisted therapy on the work engagement, burnout, pain, and quality of life among professionals working in a School for Special Education. A total of 30 participants will be involved in the program, which will be comprised of eight 50-min sessions conducted once a week. The hypothesis of the researchers in this study is that this program will achieve a reduction in burnout levels in workers, as well as an improvement in engagement and quality of life.

DETAILED DESCRIPTION:
Animal-assisted interventions have shown numerous benefits in different populations including children with cerebral palsy or autism spectrum disorder, people with chronic pain, older adults, or people in prison. Recently, different initiatives have been carried out focused on improving the work environment, especially among professionals in clinical settings and obtaining benefits in mood, as well as a reduction in the levels of stress and burnout of employees. In addition, it has also been observed that these animals in the workplace can produce an improvement in health, productivity or job satisfaction.

The presence of stress or anxiety among professionals working in Special Education Schools has been previously reported and could increase burnout and reduce the engagement and health-related quality of life of these workers.

Therefore, the current randomized controlled trial aims to evaluate the effects of an 8-week program consisting of dog-assisted therapy on the work engagement, burnout, pain, and quality of life among professionals working in a School for Special Education. A total of 30 participants will be involved in the program, which will be comprised of eight 50-min sessions conducted once a week. The hypothesis of the researchers is that this program will achieve a reduction in burnout levels in workers, as well as an improvement in engagement and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* be aged >18 years
* be workers in a School for Special Education
* work in direct contact with children (teachers, physiotherapists, etc.)

Exclusion Criteria:

* People with dog-allergy
* People with dog phobia
* People with a history of impulsive animal aggression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-26 (Estimated); Primary Completion 2021-12-23 (Estimated); Study Completion 2021-12-23 (Estimated)

PRIMARY OUTCOMES:
Changes in Burnout levels assessed using the Burnout Clinical Subtypes Questionnaire | At baseline and immediately after the intervention (within 7 days after the last session)
  The Burnout Clinical Subtypes Questionnaire (BCSQ-36) evaluates by means of 36 items the burnout of the participants. Each of the items can be scored on a Likert scale from 1 to 7; 1 being totally disagree and 7 being totally agree. In addition, the questionnaire is divided into 3 subtypes with their respective dimensions: Frantic subtype (Involvement, Ambition and Overload), Unchallenged subtype (Indifference, Boredom and Lack of Development), Worn-out subtype (Abandonment, Lack of Control and Lack of Recognition). The Burnout Clinical Subtypes Questionnaire (BCSQ-12) also assesses burnout and is calculated with the items of the BCSQ-36.
Changes in Burnout levels assessed using the Burnout Maslach Burnout Inventory (MBI) | At baseline and immediately after the intervention (within 7 days after the last session)
  The Burnout Maslach Burnout Inventory (MBI) is a tool for the assessment of burnout, as an antithesis of the UWES questionnaire focused on engagement. This questionnaire consists of 22 items that give rise to 3 dimensions: Emotional exhaustion (decrease and loss of energy or emotional resources); Depersonalization or Cynicism (negative attitudes and feelings towards the people for whom the work is intended) and Lack of personal accomplishment or professional efficacy (tendency of professionals to evaluate themselves negatively).
Changes in Burnout levels assessed using one Item for Burnout assessment | At baseline and immediately after the intervention (within 7 days after the last session)
  One Item for Burnout assessment where under the statement of "In general, according to your definition of burnout, how would you rate your level of burnout?" participants have 5 response options from "I enjoy my work. I have no symptoms of burnout" to "I feel completely burned out and often wonder if I can keep going. I am at a point where I may need some changes or should seek some kind of help."

SECONDARY OUTCOMES:
Changes in work engagement | At baseline and immediately after the intervention (within 7 days after the last session)
  Assessed through the Utrecht Work Engagement Scale (UWES), which is a scale widely used for the evaluation of engagement in the workplace . It is composed of 17 items distributed in three factors: 1) vigor (6 items, e.g., "In my work I feel full of energy"), 2) dedication (6 items, e.g., "My work has meaning") and 3) absorption (5 items, e.g., "When I am working I forget everything that happens around me"). It consists of a seven-item Likert scale (from 0 = "never" to 6 = "always").
Changes in Health-related quality of life | At baseline and immediately after the intervention (within 7 days after the last session)
  It will be assessed using the EQ-5D-5L Questionnaire (EuroQoL 5 dimensions 5 levels): it is a questionnaire consisting of 5 dimensions with 5 levels of response, the first dimension refers to mobility, the second to personal care, the third to daily activities, the fourth to pain/discomfort, and the fifth to anxiety and depression.
Changes in Health Status | At baseline and immediately after the intervention (within 7 days after the last session)
  It will be assessed using the Visual Analog Scale of the EQ-5D-5L Questionnaire (EuroQoL 5 dimensions 5 levels). It is represented as a thermometer ranging from 0 to 100, where 0 is the worst state of health that can be imagined and 100 is the best state of health imaginable.
Changes in pain | At baseline and immediately after the intervention (within 7 days after the last session)
  Assessed through a visual analog pain scale, which is represented as a thermometer ranging from 0 to 100, where 0 is the absence of pain and 100 the highest pain level imaginable
Changes in blood pressure | At baseline and immediately after the intervention (within 7 days after the last session)
  Systolic and diastolic blood pressure using the Omron MIT Elite Plus Oscillometer

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Collado-Mateo, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- King Juan Carlos University, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No